CLINICAL TRIAL: NCT04145843
Title: Registry to Evaluate the Outcomes Following Algorithmic Approach in the Endoscopic Treatment of Bile Duct Stones
Brief Title: Treatment Outcomes in Bile Duct Stones
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1504680
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Gallstone; Bile Duct Obstruction; Bile Duct Diseases
MeSH Terms: conditions — Gallstones; Cholestasis; Bile Duct Diseases | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: endoscopic retrograde cholangiopancreatography — ERCP is a procedure that enables the physician to examine the pancreatic and bile ducts and remove gallstones.
  Other Names: ERCP

SUMMARY:
This registry is to evaluate the procedural and clinical outcomes in patients undergoing endoscopic treatment of bile duct stones when utilizing an algorithmic management approach.

DETAILED DESCRIPTION:
Gallstone diseases are common, affecting 20 million patients in the United States with associated costs of over US $6 billion. Common bile duct (CBD) stones in turn occur in 15-20% patients with gallstone disease and require treatment due to risk of infection and pancreatitis. Endoscopic treatment via endoscopic retrograde cholangiopancreatography (ERCP) is the treatment modality of choice in CBD stones. The most simple treatment techniques include biliary sphincterotomy and stone extraction via the use of standard devices such as a stone retrieval balloons or stone retrieval baskets. However, patients with difficult bile duct stones require advanced maneuvers namely mechanical lithotripsy, large balloon sphincteroplasty (LBS) of the major duodenal papilla and single operator cholangioscopy-guided lithotripsy (SOC-LL).

Currently, there are no standardized treatment approaches in the management of CBD stones, especially in the management of difficult CBD stones. Therefore, ERCP in patients with difficult CBD stones can be inefficient and prolonged with use of multiple devices and techniques. In an effort to standardize the management of bile duct stones, we have devised an algorithm for the treatment of bile duct stones using current standard of care methods, taking into account the size of bile duct stones, size of bile duct and availability of endoscopic expertise. The objective of this registry is to evaluate the procedural and clinical outcomes in patients undergoing endoscopic treatment of bile duct stones when utilizing an algorithmic management approach.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with confirmed or suspected bile duct stones undergoing endoscopic therapy for treatment of bile duct stones
2. Patients 18 years or over

Exclusion Criteria:

1. Patients not undergoing endoscopic therapy for bile duct stones
2. Patients < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be selected from the patient population at the Center for interventional Endoscopy who have presented for treatment of bile duct stones.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Rate of ductal clearance at index endoscopic intervention. | 6 months
  Percent of patients that achieve ductal clearance at the index intervention

SECONDARY OUTCOMES:
Total number of needed interventions | 6 months
  Total number of endoscopic interventions required for ductal clearance
Procedure duration | Index procedure
  Length of procedure in minutes
Technical success | Index procedure
  Success of the procedures as documented by a yes or no.
Adverse Events | 6 months
  Total number of adverse events that occurred
Crossover to other therapeutic intervention | 6 months
  Need for interventional radiology or surgical intervention for bile duct stone removal as documented by yes or no.
Procedural costs | 6 months
  Total costs measured in US dollars for the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hasan, MD, Principal Investigator — AdventHealth
Locations (1):
- Center for Interventional Endoscopy, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ASGE Standards of Practice Committee; Buxbaum JL, Abbas Fehmi SM, Sultan S, Fishman DS, Qumseya BJ, Cortessis VK, Schilperoort H, Kysh L, Matsuoka L, Yachimski P, Agrawal D, Gurudu SR, Jamil LH, Jue TL, Khashab MA, Law JK, Lee JK, Naveed M, Sawhney MS, Thosani N, Yang J, Wani SB. ASGE guideline on the role of endoscopy in the evaluation and management of choledocholithiasis. Gastrointest Endosc. 2019 Jun;89(6):1075-1105.e15. doi: 10.1016/j.gie.2018.10.001. Epub 2019 Apr 9. PMID 30979521
- [Background] Ozawa N, Yasuda I, Doi S, Iwashita T, Shimizu M, Mukai T, Nakashima M, Ban T, Kojima I, Matsuda K, Matsuda M, Ishida Y, Okabe Y, Ando N, Iwata K. Prospective randomized study of endoscopic biliary stone extraction using either a basket or a balloon catheter: the BasketBall study. J Gastroenterol. 2017 May;52(5):623-630. doi: 10.1007/s00535-016-1257-2. Epub 2016 Sep 8. PMID 27631594
- [Background] Franzini T, Moura RN, Bonifacio P, Luz GO, de Souza TF, Dos Santos MEL, Rodela GL, Ide E, Herman P, Montagnini AL, D'Albuquerque LAC, Sakai P, de Moura EGH. Complex biliary stones management: cholangioscopy versus papillary large balloon dilation - a randomized controlled trial. Endosc Int Open. 2018 Feb;6(2):E131-E138. doi: 10.1055/s-0043-122493. Epub 2018 Feb 1. PMID 29399609
- [Background] Brewer Gutierrez OI, Bekkali NLH, Raijman I, Sturgess R, Sejpal DV, Aridi HD, Sherman S, Shah RJ, Kwon RS, Buxbaum JL, Zulli C, Wassef W, Adler DG, Kushnir V, Wang AY, Krishnan K, Kaul V, Tzimas D, DiMaio CJ, Ho S, Petersen B, Moon JH, Elmunzer BJ, Webster GJM, Chen YI, Dwyer LK, Inamdar S, Patrick VB, Attwell A, Hosmer A, Ko C, Maurano A, Sarkar A, Taylor LJ, Gregory MH, Strand DS, Raza A, Kothari S, Harris JP, Kumta NA, Manvar A, Topazian MD, Lee YN, Spiceland CM, Trindade AJ, Bukhari MA, Sanaei O, Ngamruengphong S, Khashab MA. Efficacy and Safety of Digital Single-Operator Cholangioscopy for Difficult Biliary Stones. Clin Gastroenterol Hepatol. 2018 Jun;16(6):918-926.e1. doi: 10.1016/j.cgh.2017.10.017. Epub 2017 Oct 24. PMID 29074446
- [Background] Aburajab M, Dua K. Endoscopic Management of Difficult Bile Duct Stones. Curr Gastroenterol Rep. 2018 Mar 23;20(2):8. doi: 10.1007/s11894-018-0613-1. PMID 29572696
- [Background] Cote GA, Singh S, Bucksot LG, Lazzell-Pannell L, Schmidt SE, Fogel E, McHenry L, Watkins J, Lehman G, Sherman S. Association between volume of endoscopic retrograde cholangiopancreatography at an academic medical center and use of pancreatobiliary therapy. Clin Gastroenterol Hepatol. 2012 Aug;10(8):920-4. doi: 10.1016/j.cgh.2012.02.019. Epub 2012 Mar 2. PMID 22387254
- [Background] Rosenkranz L, Patel SN. Endoscopic retrograde cholangiopancreatography for stone burden in the bile and pancreatic ducts. Gastrointest Endosc Clin N Am. 2012 Jul;22(3):435-50. doi: 10.1016/j.giec.2012.05.007. Epub 2012 Jun 12. PMID 22748241
- [Background] Karsenti D, Coron E, Vanbiervliet G, Privat J, Kull E, Bichard P, Perrot B, Quentin V, Duriez A, Cholet F, Subtil C, Duchmann JC, Lefort C, Hudziak H, Koch S, Granval P, Lecleire S, Charachon A, Barange K, Cesbron EM, De Widerspach A, Le Baleur Y, Barthet M, Poincloux L. Complete endoscopic sphincterotomy with vs. without large-balloon dilation for the removal of large bile duct stones: randomized multicenter study. Endoscopy. 2017 Oct;49(10):968-976. doi: 10.1055/s-0043-114411. Epub 2017 Jul 28. PMID 28753698
- [Background] Buxbaum J, Sahakian A, Ko C, Jayaram P, Lane C, Yu CY, Kankotia R, Laine L. Randomized trial of cholangioscopy-guided laser lithotripsy versus conventional therapy for large bile duct stones (with videos). Gastrointest Endosc. 2018 Apr;87(4):1050-1060. doi: 10.1016/j.gie.2017.08.021. Epub 2017 Sep 1. PMID 28866457
- [Background] Varadarajulu S, Kilgore ML, Wilcox CM, Eloubeidi MA. Relationship among hospital ERCP volume, length of stay, and technical outcomes. Gastrointest Endosc. 2006 Sep;64(3):338-47. doi: 10.1016/j.gie.2005.05.016. PMID 16923479